CLINICAL TRIAL: NCT07324187
Title: Peri-implant Soft Tissue Thickness in the Aesthetic Zone: A Randomized Controlled Clinical Trial Comparing Connective Tissue Grafts and a Volume-Stable Collagen Matrix
Brief Title: CTG vs VCMX for Peri-implant Soft Tissue Thickness
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical Innovation Center Wroclaw (Other)
Collaborators: Geistlich Pharma AG (Industry)
Responsible Party: Principal Investigator, Jakub Hadzik, Associate Professor, PhD, DSc (Med.), Specialist in Oral Surgery, Medical Innovation Center Wroclaw
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 400166
Record Dates: First submitted 2025-12-23; First posted 2026-01-07 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2025-12

CONDITIONS: Dental Implants; Peri-Implant Tissues; Missing Tooth/Teeth
Keywords: connective tissue graft,; collagen matrix; peri-implant soft tissue; CTG; VCMX
MeSH Terms: conditions — Anodontia

STUDY DESIGN:
Intervention Model Description: Participants were randomly assigned in a 1:1 ratio to one of two parallel intervention groups.
Who Masked: Outcomes Assessor
Masking Description: Clinical outcome assessments were performed by an independent examiner who not involved in the surgical procedures unaware of group allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Connective Tissue Graft (CTG) (Active Comparator): Participants received peri-implant soft tissue augmentation using an autogenous subepithelial connective tissue graft harvested from the palate and placed at the implant site according to a standardized surgical protocol.
  Interventions: Procedure: Connective Tissue Graft
- Volume-Stable Collagen Matrix (VCMX) (Experimental): Participants received peri-implant soft tissue augmentation using a volume-stable collagen matrix placed at the implant site according to the manufacturer's instructions and a standardized surgical protocol.
  Interventions: Device: Volume-Stable Collagen Matrix

INTERVENTIONS:
Procedure: Connective Tissue Graft — An autogenous subepithelial connective tissue graft harvested from the palatal donor site and used for peri-implant soft tissue augmentation according to a standardized surgical protocol.
  Arms: Connective Tissue Graft (CTG)
Device: Volume-Stable Collagen Matrix — A volume-stable collagen matrix used for peri-implant soft tissue augmentation according to the manufacturer's instructions and a standardized surgical protocol.
  Arms: Volume-Stable Collagen Matrix (VCMX)

SUMMARY:
This investigator-initiated randomized controlled clinical trial evaluated changes in peri-implant soft tissue thickness in the aesthetic zone following soft tissue augmentation. Adult patients requiring single-tooth implant therapy in the aesthetic zone were randomly assigned to receive either an autogenous connective tissue graft (CTG) or a volume-stable collagen matrix (VCMX) at the implant site.

The primary objective of the study was to compare changes in peri-implant soft tissue thickness between the two treatment approaches over time. Secondary objectives included evaluation of aesthetic outcomes, clinical parameters, and treatment-related complications.

The study was conducted at a single academic clinical center in Poland in accordance with Good Clinical Practice, the Declaration of Helsinki, and applicable ethical and regulatory requirements. All participants provided written informed consent prior to enrollment.

DETAILED DESCRIPTION:
This investigator-initiated, single-center, randomized controlled clinical trial was designed to assess the effectiveness of two different soft tissue augmentation approaches on peri-implant soft tissue thickness in the aesthetic zone. The study compared the use of an autogenous connective tissue graft (CTG) with a volume-stable collagen matrix (VCMX) in patients undergoing single-tooth implant therapy.

Eligible adult patients presenting with an indication for peri-implant soft tissue augmentation in the aesthetic zone were enrolled and randomly allocated in a 1:1 ratio to one of the two intervention groups. In the CTG group, a subepithelial connective tissue graft was harvested from the palate and placed at the peri-implant site. In the VCMX group, a commercially available volume-stable collagen matrix was used for soft tissue augmentation according to the manufacturer's instructions.

Standardized surgical and prosthetic protocols were applied in both groups. Clinical examinations and outcome assessments were performed at predefined follow-up visits. The primary outcome measure was the change in peri-implant soft tissue thickness measured at the implant site over time. Secondary outcome measures included additional clinical parameters, aesthetic outcomes, patient-reported outcomes, and the incidence of adverse events or complications.

The study protocol, patient information sheet, and informed consent form were approved by the Bioethics Committee of Wroclaw Medical University prior to study initiation. The study was conducted in compliance with Good Clinical Practice guidelines, ISO 14155, and the principles of the Declaration of Helsinki. All participants provided written informed consent before any study-related procedures were performed.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 years or older.
* Single-tooth edentulism in the aesthetic zone of the maxilla or mandible, bordered by natural teeth on both sides.
* Bilateral two-tooth edentulism accepted only when implants were placed in separate quadrants.
* Indication for dental implant placement with peri-implant soft tissue augmentation.
* Adequate bone volume at the implant site confirmed radiographically.
* Baseline peri-implant soft tissue thickness suitable for augmentation.
* Minimum height of keratinized tissue of at least 2 mm.
* Good oral hygiene and periodontal health.
* Ability and willingness to provide written informed consent.

Exclusion Criteria:

* Previous bone grafting procedures at the intended implant site.
* Severe periodontal disease or untreated oral infection.
* Bruxism or heavy smoking.
* Systemic diseases or conditions that could impair wound healing or bone metabolism.
* History of radiotherapy in the head and neck region.
* Previous or ongoing bisphosphonate therapy.
* Uncontrolled diabetes mellitus.
* Pregnancy or breastfeeding.
* Use of medications known to interfere with soft tissue healing.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2022-01-02 (Actual); Primary Completion 2025-04-10 (Actual); Study Completion 2025-04-19 (Actual)

PRIMARY OUTCOMES:
Change in peri-implant soft tissue thickness | Baseline and 6 months after soft tissue augmentation
  Change in peri-implant soft tissue thickness measured at the implant site using a standardized clinical measurement method.

SECONDARY OUTCOMES:
Peri-implant soft tissue thickness at additional follow-up time points | Baseline, 3 months, and 12 months after augmentation
  Peri-implant soft tissue thickness assessed at predefined follow-up visits after soft tissue augmentation.

CONTACTS AND LOCATIONS:
Locations (1):
- Medyczne Centrum Innowacji Wrocław (Wrocław Medical Innovation Center), formerly operating as Akademicka Akademicka Poliklinika Stomatologiczna, Wroclaw, Poland

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared due to data protection and confidentiality considerations, and because informed consent for public data sharing was not obtained from participants.